CLINICAL TRIAL: NCT06525948
Title: Efficacy and Safety of rhTPO in Combination With Cyclosporine Versus Cyclosporine Alone in the Treatment of Transfusion-dependent Non-severe Aplastic Anaemia (TD-NSAA)
Brief Title: Efficacy and Safety of rhTPO in Combination With Cyclosporine Versus Cyclosporine Alone in the Treatment of TD-NSAA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, chief physician, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rTC-AA
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Aplastic Anemia; Transfusion-dependent Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- two-drug combination group (Experimental): rhTPO combined with cyclosporine
  Interventions: Drug: rhTPO; Drug: Cyclosporin A
- drug-free group (Active Comparator): cyclosporine alone
  Interventions: Drug: Cyclosporin A

INTERVENTIONS:
Drug: rhTPO — rhTPO
  Arms: two-drug combination group
Drug: Cyclosporin A — cyclosporine A

SUMMARY:
Investigating the efficacy and safety of rhTPO in combination with cyclosporine versus cyclosporine alone for the treatment of TD-NSAA

DETAILED DESCRIPTION:
Investigating the efficacy and safety of rhTPO in combination with cyclosporine versus cyclosporine alone for the treatment of transfusion-dependent aplastic anaemia of the non-severe type

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥ 18 years, male and female; 2. patients with a clear diagnosis of NSAA who are dependent on transfusion therapy:

1. Meet the Camitta NSAA criteria;
2. accompanied by at least one of the following abnormalities: (1) dependence on component blood transfusion therapy, at least one component blood transfusion every 8 weeks on average, and the duration of transfusion dependence ≥ 4 months, the indication of component blood transfusion: HGB ≤ 60g / L; (2) PLT ≤ 10 × 10 ^ 9 / L, or PLT ≤ 30 × 10 ^ 9 / L with a significant tendency to bleed; (3) neutrophils ≤ 0.5 × 10 ^ 9 / L.
3. Excluding other haematological and non-haematological diseases that cause pancytopenia; 3. ECOG PS score 0-2, expected survival ≥ 3 months with follow-up; 4. functional levels of major organs must meet the following requirements: 1) Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); 2) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN; 3) blood creatinine (Cr) ≤ 1.5 x ULN; 5. has not been treated with platelet receptor agonist (TPO-RA) analogues and other immunosuppressant analogues; 6. the subject is not suitable or willing to receive haematopoietic stem cell transplantation therapy; 7. no history of serious heart, lung, liver, kidney and other important organs and endocrine system diseases; 8. Voluntarily enroll in the study, sign the informed consent, have good compliance and willing to cooperate with the follow-up.

Exclusion Criteria:

1. have used other clinical investigational drugs within 4 weeks;
2. a history of primary myelodysplastic syndromes (MDS), primary paroxysmal sleep haemoglobinuria (PNH) and leukaemia, as well as congenital bone marrow failure syndromes (IBMFS), such as Fanconi's anaemia (FA) and congenital dyskeratosis (DC)
3. history of cirrhosis or history of portal hypertension;
4. congestive heart failure, arrhythmia, peripheral arteriovenous thrombosis requiring medication within 1 year prior to enrolment, or myocardial infarction or cerebral infarction within 3 months prior to enrolment;
5. HIV infection;
6. severe autoimmune disease or immunodeficiency disease;
7. suffering from malignant tumour
8. severe mental disorders;
9. a known history of allergy to the drug components of this regimen;
10. in the opinion of the investigator, it is not appropriate to participate in this trial, e.g., any other medical, social or psychological factors that may affect safety or compliance with the study procedures.

Compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 months
  Overall Response Rate (ORR): meets the criteria for CR and PR.
CRR | 3 months
  Complete Response Rate (CRR)：ANC>1.5×10^9/L，Hb>100g/L，PLT>100×10^9/L；

SECONDARY OUTCOMES:
ORR | 6 months
  Overall Response Rate (ORR): meets the criteria for CR and PR.
CRR | 6 months
  Complete Response Rate (CRR)：ANC>1.5×10^9/L，Hb>100g/L，PLT>100×10^9/L；
Time for platelet count to recover to ≥20 x 10^9/L with a 1-fold increase in absolute value | through study completion, an average of 1 year
  Time for platelet count to recover to ≥20 x 10^9/L with a 1-fold increase in absolute
Proportion of patients with adverse events | through study completion, an average of 1 year
  safety event

CONTACTS AND LOCATIONS:
Overall Officials: Bing Han, PhD, Principal Investigator — Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young NS. Aplastic anaemia. Lancet. 1995 Jul 22;346(8969):228-32. doi: 10.1016/s0140-6736(95)91273-8. No abstract available. PMID 7616805
- [Background] Dancan GD. Spectrophotometry of tissue glycogen. Clin Chem. 1984 Sep;30(9):1580-1. No abstract available. PMID 6467577
- [Background] Bacigalupo A. How I treat acquired aplastic anemia. Blood. 2017 Mar 16;129(11):1428-1436. doi: 10.1182/blood-2016-08-693481. Epub 2017 Jan 17. PMID 28096088
- [Background] Yang C, Zhang X. Incidence survey of aplastic anemia in China. Chin Med Sci J. 1991 Dec;6(4):203-7. PMID 1813058